CLINICAL TRIAL: NCT00692588
Title: Magnetic Resonance Imaging to Measure Treatment Effects of Doxycycline and Rifampicin in Alzheimer's Disease
Brief Title: MRI to Measure Treatment With Antibiotics in Alzheimer's Disease
Acronym: DARAD-MRI
Status: Completed | Type: Observational
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: St. Peter's Hospital (Unknown); St. Peter's Centre for Studies in Aging (Unknown)
Responsible Party: Dr. Mohammed Ali Warsi, McMaster University
Other Study IDs: R.P. #07-2949
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Diffusion Tensor Imaging; Susceptibility Weighted Imaging; Doxycycline; Rifampicin
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Placebo: Subjects who received placebo in DARAD Trial
- Doxycycline: Subjects who received doxycycline in DARAD Trial
- Rifampicin: Subjects who received rifampicin in DARAD Trial
- Doxycycline and Rifampicin: Subjects who received doxycycline and rifampicin in DARAD Trial
- Control: Normal controls

SUMMARY:
Objectives:

To study the changes in brain structure and function using MRI scans in patients treated for Alzheimer's disease.

Methods:

A pilot study of treating Alzheimer's disease with antibiotics showed some promise that this treatment could delay the deterioration of the mind with this disease. This study is being replicated on a larger scale, providing a more definitive answer to this question. In addition to looking at changes of the mind (through cognitive tests), we would like to use MRI scans in these patients before and after treatment to study the structural changes and the chemical changes in the brain. This would provide a non-invasive look at the bran processes that protect the brain from the effect of Alzheimer's as well as confirming that the disease has been modified with treatment.

Impact:

The novel treatment of Alzheimer's with antibiotics has provided a potential breakthrough in the field. In addition to verifying changes in the brain, MRI scans can observe HOW this process could occur, thus opening doors to other new treatments for Alzheimer's and perhaps even cures.

ELIGIBILITY:
Inclusion Criteria:

(DARAD Trial)

1. Male or female aged 50 years or older.
2. Diagnosis of dementia using standardized DSM IV criteria and probable Alzheimer's disease (NINCDS-ADRDA criteria).
3. SMMSE score 14-26 inclusive.
4. Patients who have a consistent caregiver who will accompany them to clinic visits, ensure medication compliance, monitor and report adverse events and sign informed consent for his or her own participation.
5. Sufficient visual, hearing and communication skills to complete standardized testing in English.
6. Patients or their legally acceptable representatives for personal care who sign informed consent.
7. Otherwise healthy on physical examination and screening physical and laboratory testing.

Exclusion Criteria:

(DARAD Trial)

1. Patients with neurodegenerative diseases such as Lewy Body dementia, Parkinson's disease, Fronto-temporal Dementia, Huntington's Chorea, Down's Syndrome or Creutzfeld Jacob Disease.
2. Cognitive impairment which may be due to any of the following conditions:

   1. acute cerebral trauma, subdural hematoma, injuries from chronic trauma like boxing.
   2. Hypoxic cerebral damage e.g. post cardiac arrest, postanesthesia etc.
   3. Vitamin deficiency like B12 deficiency will be treated and stabilized for one month before patients will be randomized to the study. Patients taking B12 for more than one month can be included in the study.
   4. Infections like cerebral abscesses, herpes, neurosyphilis, meningitis or AIDS.
   5. Primary or metastatic cerebral neoplasia.
   6. Endocrine deficiencies like hypercalcemia, hypothyroidism, hyperparathyroidism, Cushing's syndrome, severe renal failure, poorly controlled diabetes mellitus, pituitary disease, etc.
   7. Mental retardation. If a patient has one of these conditions and in the opinion of the investigator this condition has stabilized and is not contributing to the decline in cognition then this patient may be included in the study after the steering committee has reviewed the situation and approved participation.
3. Multi-infarct dementia or significant cerebrovascular disease as evidenced by a) stroke with deficit that may confound the assessment of cognitive function or b) multiple focal signs on exam indicative of multiple ischemic events or c) findings on CT or MRI scan that show multiple lacunar infarcts, extensive periventricular white matter lesion, an infarct in the angular gyrus, the thalamus, the basal forebrain, the anterior or posterior cerebral artery territory.
4. Patients with significant intracranial pathology such as tumour or hydrocephalus confirmed by CT or MRI in the past two years. The CT or MRI must be repeated before inclusion if the patient has experienced significant loss of consciousness or other neurological signs or symptoms, step-wise deterioration or has sustained a significant head injury since the last scan was performed. Patients with loss of consciousness, transient ischemic attacks or drop attacks, may be considered if these did not occur in the preceding twelve months.
5. Patients with the following co-existing medical conditions:

   1. History of epilepsy or convulsions.
   2. Clinically significant psychiatric conditions (based on DSM-IV criteria) like major depression, schizophrenia. A Cornell Scale for Depression in Dementia score of 12 or more out of 38.
   3. Moderate to severe behavioural disturbances,
   4. Clinically significant hepatic, renal, pulmonary, metabolic or endocrine diseases.
   5. History of drug or alcohol abuse in the year prior to enrolment.
   6. History of myasthenia gravis.
6. Clinically significant cardiac disease such as:

   1. Cardiac surgery in the past six months.
   2. Unstable angina or poorly controlled congestive heart failure (NYHA III or IV).
   3. Uncontrolled hypertension with systolic pressure greater that 180 mmHg. or diastolic pressure greater that 110 mmHg.
7. Patients taking anti-dementia treatments with the following exceptions: donepezil, galantamine, rivastigmine, memantine, ASA up to 650 mg OD, Vitamin E 400 i.u., multi B vitamins, Ginko biloba, Cox II inhibitors or statins. In all cases the dose should have been stable for three months or more, and not be expected to change for the duration of the trial.
8. Patients enrolled in other clinical trials with investigational drugs.
9. Patients taking long term antibiotics (more than one month in the past six months).
10. Allergies to these antibiotics.

(MRI)

1. Cardiac pacemaker or implantable defibrillator
2. Cerebral aneurysm clip
3. Neural stimulator (e.g. TENS-Unit)
4. Any type of ear implant
5. Ocular foreign body (e.g. metal shavings)
6. Any implanted device (e.g. insulin pump, drug infusion device)
7. Metal shrapnel or bullet.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in the DARAD Trial (Doxycycline and Rifampicin for Alzheimer's disease).
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Changes in MRI Pre Vs Post Treatment | 1 Year

SECONDARY OUTCOMES:
Comparison of Normal Controls Vs Alzheimer's Disease using MRI | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Warsi, (Hon)BSc, MSc, MD, FRCP(C), Principal Investigator — McMaster University; Michael D Noseworthy, (Hon)BSc, MSc, PhD, Study Director — St. Joseph's Hospital; William Molloy, MBBch, MRCP, FRCP(C), Study Director — St. Peters Hospital
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada